CLINICAL TRIAL: NCT02426853
Title: Sun Protection, Tanning Behaviors and Attitudes in Adolescents
Brief Title: Ultraviolet (UV) Photography in Adolescents
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014-1037; NCI-2015-00764 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-04-22; First posted 2015-04-27 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Cancer Prevention
Keywords: Cancer Prevention; Sun protection; Photograph; UV photograph; Ultraviolet; Pamphlets; Handouts; Questionnaires; Surveys; Skin cancer risk behaviors
MeSH Terms: interventions — Surveys and Questionnaires; Motion Pictures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - UV Photography Group (Experimental): Participants complete 1 questionnaire at beginning of study, 1 after receiving education about how to protect skin from sun and how to avoid tanning beds, and 1 at about 3 months after receiving skin protection education. Participants given handouts that discusses skin cancer prevention, sun protection, and how to avoid tanning beds. At beginning of study, 2 photos taken of the face. One photo is a standard photo, the other photo is taken with an ultraviolet (UV) filter.
  Interventions: Behavioral: Questionnaires; Other: Photos; Behavioral: Pamphlets
- Group 2 - Comparison Group (Active Comparator): Participants complete 1 questionnaire at beginning of study, 1 after receiving education about how to protect skin from sun and how to avoid tanning beds, and 1 at about 3 months after receiving skin protection education. Participants given handouts that discusses skin cancer prevention, sun protection, and how to avoid tanning beds.
  Interventions: Behavioral: Questionnaires; Behavioral: Pamphlets

INTERVENTIONS:
Behavioral: Questionnaires — Participants complete 1 questionnaire at beginning of study, 1 after receiving education about how to protect skin from sun and how to avoid tanning beds, and 1 at about 3 months after receiving skin protection education.
  Other Names: Surveys
Other: Photos — At beginning of study, 2 photos taken of the face. One photo is a standard photo, the other photo is taken with an ultraviolet (UV) filter.
  Other Names: Pictures
  Arms: Group 1 - UV Photography Group
Behavioral: Pamphlets — At beginning of study, handouts given that discusses skin cancer prevention, sun protection, and how to avoid tanning beds.
  Other Names: Handouts

SUMMARY:
The goal of this research study is to learn how students react to seeing a photograph of any skin damage they may have on their face. This skin damage may be caused by sun exposure or use of tanning beds. Researchers also want to learn about students' sun protection, tanning behaviors, and attitudes towards sun exposure, sun protection, tanning behaviors and skin cancer.

Researchers will use the results of this study to design programs for students about sun protection and tanning avoidance.

DETAILED DESCRIPTION:
If participant agrees to take part in this study, they will complete 3 questionnaires about sun protection, tanning behaviors, sunburns, and attitudes and opinions about sun exposure, sun protection, tanning behaviors and skin cancer.

Participant's school will be assigned to 1 of 2 possible groups:

* If participant's school is assigned to Group 1, they will have 2 photos taken of their face. One (1) photo is a standard photo (like the kind one may take with a regular camera). The other photo is taken with an ultraviolet (UV) filter and shows skin damage that cannot be seen in a standard photo.
* If participant's school is assigned to Group 2, they will not have any photos taken.

If participant is in Group 1, they and a member of the study staff will compare the standard and UV photographs together. The study staff will discuss any skin damage seen with participant. A member of the study staff will record on a paper form any visible reactions participant may have to viewing their UV photograph. Participant will also be given a handout that discusses skin cancer prevention, sun protection, and how to avoid tanning beds. Participant will see their photos on a computer screen. Participant will not be given their photos. At the end of this study, the photos will be deleted.

If participant is in Group 2, they will only receive a handout that discusses skin cancer prevention, sun protection, and how to avoid tanning beds.

All participants will complete 1 questionnaire at the beginning of the study (before receiving any kind of education about skin cancer prevention), 1 questionnaire after receiving education about how to protect participant's skin from the sun and how to avoid tanning beds, and 1 questionnaire at about 3 months after receiving the education about how to protect skin from the sun and how to avoid tanning beds.

Participant will complete these study procedures at school and they may answer some of the questionnaires outside of school. Participant will complete the first questionnaire on paper at their school. Participant will have an option to complete this questionnaire online if they are not able to complete it on paper the day the study team visits their school. Participant will complete the second questionnaire on paper at their school. Participant will complete the third questionnaire online. Links to the online questionnaires will be sent to the email address that participant will provide on the Participant Contact Information Form. Participant will also have an option to receive a link to the questionnaire via text message if they provide us with a cell phone number that can receive text messages on the Participant Contact Information Form. Participant may incur charges for receiving text messages.

Length of Study:

Student's participation in this study will be over after they have completed the last questionnaire. It will take about 1 hour to complete all study questionnaires and procedures.

This is an investigational study.

Up to 420 participants will be enrolled in this study. All will take part through MD Anderson at different schools in the greater Houston area.

Only about 35 participants will be able to take part at each school. This means that even if participant agrees, they may not be selected to take part in this study. The student participants will be randomly selected from the pool of students who agree to participate.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in 7th or 8th grade
2. Ability to speak, read and write English
3. Has email address and internet access to complete online surveys
4. Willingness to provide contact information including phone number, email address and mailing address

Exclusion Criteria:

1) N/A

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 293 (Actual)
Dates: Start 2015-04-21 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
Sun Protection Behavior Composite Score | 3 months
  Baseline sun protection behaviors are assessed using self-reported measures of sun protection behaviors. Both the baseline and 3-month behavior composite scores range from 1 to 5 and are calculated as the mean of the four sun protection behavior items.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Peterson, MPH,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- Houston Independent School District, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org